CLINICAL TRIAL: NCT06721806
Title: Role of Platelet Rich Plasma in Bone Regeneration After Enucleation of Odontogenic Jaw Cysts
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maikel Merit Gerges Morkos, resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRP & bone healing
Record Dates: First submitted 2024-11-05; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: PRP & Jaw Cysts
MeSH Terms: conditions — Jaw Cysts | interventions — Bone Regeneration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP and bone regeneration after enucleation of odontogenic jaw cysts (Active Comparator): effect of PRP on regeneration
  Interventions: Procedure: PRP & bone regeneration
- bone regeneration power without PRP (Placebo Comparator): bone healing without use of PRP
  Interventions: Procedure: PRP & bone regeneration

INTERVENTIONS:
Procedure: PRP & bone regeneration — PRP effect on bone healing

SUMMARY:
in the present study, the effect of PRP on bone regeneration when applied to the site of removal of cyst of the jaws is evaluated. PRP was delivered to the site combined with gelfoam. Thrombin clot accelerator was not used.

DETAILED DESCRIPTION:
Jaw cysts are common lesions in the oral and maxillofacial region. Enucleation of cyst wall & curettage has evolved as the treatment of choice. In order to reduce infections and to accelerate bone regeneration, by using of Platelet rich plasma.

Platelets are involved in regeneration at sites of pathology, apart from their role in clotting. A preparation composed mainly of platelets (platelet-rich plasma gel) applied to sites of bony pathology, after surgical treatment of lesions, may hasten bone regeneration.

An interesting idea developed that the addition of a concentrate of platelets, to wounded tissues or surgical sites, may enhance the body's natural wound healing mechanisms . Platelet-rich plasma (PRP) is the accepted term to describe the preparation made out of autologous platelets suspended in autologous plasma, in concentration greater than normally found in peripheral blood Because it is autologous, PRP avoids the risk of transmissible diseases such as HIV, Hepatitis B, C or D and other blood-borne pathogens .A clot accelerator such as bovine thrombin is added to gel the PRP or PRP is added to other materials such as collagen, gelfoam, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Size of the cyst more than 2 cm
2. The lesion could be visualized radiographically
3. Patients within the age range of 20 to 50 years

Exclusion Criteria:

1. Patients who were alcoholics & smokers
2. -Patients with systemic diseases
3. History of bleeding tendencies, blood dyscrasia
4. Low platelet count
5. Patients unable or unwilling to return for follow-up

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
bone healing | 6 months
  effect of PRP in bone healing by measuring bone density
PRP & infection rate | 6 months
  PRP reduce infection rate

REFERENCES:
- [Background] Tiwari A. A Traumatic Ulcer Caused by Accidental Lip Biting Following Topical Anesthesia: A Case Report. Cureus. 2023 Apr 29;15(4):e38316. doi: 10.7759/cureus.38316. eCollection 2023 Apr. PMID 37261171
- [Background] Dohan DM, Choukroun J, Diss A, Dohan SL, Dohan AJ, Mouhyi J, Gogly B. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part I: technological concepts and evolution. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e37-44. doi: 10.1016/j.tripleo.2005.07.008. Epub 2006 Jan 19. PMID 16504849
- [Background] Dohan DM, Choukroun J, Diss A, Dohan SL, Dohan AJ, Mouhyi J, Gogly B. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part II: platelet-related biologic features. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e45-50. doi: 10.1016/j.tripleo.2005.07.009. Epub 2006 Jan 10. PMID 16504850
- [Background] Intini G. The use of platelet-rich plasma in bone reconstruction therapy. Biomaterials. 2009 Oct;30(28):4956-66. doi: 10.1016/j.biomaterials.2009.05.055. Epub 2009 Jul 1. PMID 19573909
- [Background] Rathore A, Tiwari A, Nazim M, Gupta AK, Gande M, Krishnakumar J. Detection of Human PapillomaVirus and its Association with Potentially Malignant Disorders and Oral Squamous Cell Carcinoma: A Retrospective Study. J Pharm Bioallied Sci. 2022 Jul;14(Suppl 1):S820-S824. doi: 10.4103/jpbs.jpbs_9_22. Epub 2022 Jul 13. PMID 36110657
- [Background] Raghavendra KM, Sara TB, Mariam VJ, Bhat GS. Author's reply: Platelet-rich fibrin as an adjunct to palatal wound healing after harvesting a free gingival graft: A case series. J Indian Soc Periodontol. 2014 Nov-Dec;18(6):684-5. doi: 10.4103/0972-124X.147397. No abstract available. PMID 25624621
- [Background] Kulkarni MR, Thomas BS, Varghese JM, Bhat GS. Platelet-rich fibrin as an adjunct to palatal wound healing after harvesting a free gingival graft: A case series. J Indian Soc Periodontol. 2014 May;18(3):399-402. doi: 10.4103/0972-124X.134591. PMID 25024559

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-11-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT06721806/Prot_SAP_ICF_000.pdf